CLINICAL TRIAL: NCT05026736
Title: A Phase 2 Clinical Trial Evaluating the Efficacy and Safety of Sintilimab for Angiosarcoma
Brief Title: Sintilimab for the Treatment of Locally Advanced, Metastatic, or Recurrent Angiosarcoma, the SiARa Cancer Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI request, <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1212; NCI-2021-08962 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1212 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Angiosarcoma; Metastatic Angiosarcoma; Recurrent Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sintilimab) (Experimental): Patients receive sintilimab IV over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may continue to receive treatment at the discretion of the treating physician.
  Interventions: Other: Quality-of-Life Assessment; Biological: Sintilimab

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Sintilimab — Given IV
  Other Names: Anti-PD-1 Monoclonal Antibody IBI308; Anti-PDCD1 Monoclonal Antibody IBI308; IBI 308; IBI308

SUMMARY:
This phase II trial evaluates the effect of sintilimab in treating patients with angiosarcoma that has spread to nearby tissue or lymph nodes (locally advanced), has spread to other places in the body (metastatic), or has come back (recurrent). Immunotherapy with monoclonal antibodies, such as sintilimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving sintilimab may help to control angiosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of sintilimab in subjects with angiosarcoma (progression- free rate PFR at 9 cycles by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).

SECONDARY OBJECTIVE:

I. To evaluate the objective response rate (ORR), stable disease rate (SDR), progression free survival (PFS), overall survival (OS), quality of life (QOL), safety and duration of response (DOR) of sintilimab in subjects with angiosarcoma.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation between biomarkers in tumor tissue and efficacy, including but not restricted to PD-L1 expression level, transcriptome sequencing, single-cell sequencing, and multicolor immunohistochemistry (IHC) analyses.

II. To evaluate the correlation between biomarkers in peripheral blood and efficacy, including but not restricted to soluble PD-L1, circulating tumor deoxyribonucleic acid (DNA) (ctDNA), and cytokine analyses.

OUTLINE:

Patients receive sintilimab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may continue to receive treatment at the discretion of the treating physician.

After completion of study treatment, patients are followed up at 30 and 90 days, and then every 60 days for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed unresectable, locally advanced, recurrent or metastatic angiosarcoma
* Intolerant to or progressed on at least one line of systemic chemotherapy. Patient ineligible for cytotoxic chemotherapy are eligible
* Aged >= 18
* Can provide archival or fresh tissues for optional correlative analysis
* Have at least one measurable lesion as per RECIST version (v)1.1
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet (PLT) count >= 75 x 10^9/L
* Hemoglobin (HGB) >= 8.0 g/dL
* Total bilirubin (TBIL) =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN in subjects without hepatic metastasis; ALT and AST =< 5 x ULN in subjects with hepatic metastasis, gamma-glutamyl transferase (GGT) =< 10 x ULN
* Urine protein < 2+ from random sample or < 1 g from 24-hour urine collection
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance rate (Ccr) >= 50 mL/min by Cockcroft-Gault formula
* Adequate coagulation function, defined as international normalized ratio (INR) =< 1.5 or prothrombin time (PT) =< 1.5 x ULN; if the subject is receiving anticoagulant therapy, the results of coagulation tests need to be within the acceptable range for anticoagulants
* Expected survival >= 12 weeks
* Subject (female subjects of childbearing age or male subjects whose partners are of childbearing age) must take effective contraceptive measures during the entire course of the trial and until 180 days after the last dose
* Signed the informed consent form (ICF) and be able to comply with the scheduled follow-up visits and related procedures required in the protocol

Exclusion Criteria:

* Received treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug that specifically targets T-cell co-stimulation or immune checkpoint pathways
* Enrolled in another interventional clinical study for angiosarcoma, unless only involved in an observational study (non-interventional) or in the follow-up phase of an interventional study
* Received palliative radiation therapy for local lesion within 2 weeks prior to the first dose
* Received systemic treatment with anti-cancer indications or immunomodulators (including thymosins, interferons, and interleukins) within 2 weeks prior to the first dose of study treatment
* Received systemic immunosuppressants within 2 weeks prior to first dose, excluding local use of glucocorticoids administered by nasal, inhaled, or other routes, and systemic glucocorticoids at physiological doses (no more than 10 mg/day of prednisone or equivalents), or glucocorticoids to prevent allergies to contrast media
* Received a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or be scheduled to receive live attenuated vaccine during the study period

  * Note: Seasonal inactivated influenza virus vaccines within 4 weeks prior to the first dose of study treatment are permitted, but attenuated influenza vaccines are not
* Received major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or is scheduled to receive major surgery during the course of the trial
* Any toxicity (excluding alopecia, events that are not clinically significant, or asymptomatic laboratory abnormalities) due to prior anti-tumor therapy that has not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 grade 0 or 1 prior to the first dose of study treatment
* Known symptomatic central nervous system (CNS) metastasis or carcinomatous meningitis. Subjects with brain metastases who have received prior treatment can be enrolled if the disease is stable (no imaging evidence of progressive disease [PD] for at least 4 weeks prior to the first dose of study treatment), there is no evidence of new brain metastases or progression of the existing metastatic lesion(s) upon repeated imaging, and corticosteroids have not been required for at least 14 days prior to the first dose of study treatment. Patients with carcinomatous meningitis are ineligible, regardless of whether the disease is clinically stable or not
* Subjects with bone metastases at risk of paraplegia
* Known active autoimmune disease requiring treatment or previous disease history within 2 years (subjects with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment, hypothyroidism only requiring thyroid replacement, or type I diabetes only requiring insulin can be enrolled)
* Known history of primary immunodeficiency diseases
* Known active pulmonary tuberculosis
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Human immunodeficiency virus (HIV)-infected subjects (positive anti-HIV antibody)
* Active or poorly controlled serious infections that require systemic therapy
* Symptomatic congestive heart failure (New York Heart Association [NYHA] class II-IV) or symptomatic or poorly controlled arrhythmia
* Uncontrolled hypertension (systolic blood pressure >= 160 mmHg or diastolic blood pressure >= 100 mmHg) despite of standard treatment
* Any arterial thromboembolic event within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack
* Significant malnutrition, such as those requiring continuous parenteral nutrition >= 7 days; excluding those having received intravenous treatment for malnutrition for more than 4 weeks before the first dose of study treatment
* History of clinically significant deep venous thrombosis, pulmonary embolism, or other serious thromboembolic events within 3 months prior to enrollment (implantable port or catheter-related thrombosis or incidental pulmonary embolism [PE] detected on scan without symptoms or superficial venous thrombosis are not considered as "serious" thromboembolisms)
* Uncontrolled metabolic disorders, non-malignant organ or systemic diseases, or cancer-related secondary diseases that may lead to higher medical risks and/or survival evaluation uncertainties
* Hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh class B or C
* Bowel obstruction or history of the following diseases: inflammatory bowel disease, extensive bowel resection (partial colectomy or extensive small intestine resection accompanied with chronic diarrhea), Crohn's disease, or ulcerative colitis
* Known acute or chronic active hepatitis B (positive hepatitis B surface antigen [HBsAg] and hepatitis B virus [HBV] deoxyribonucleic acid [DNA] viral load >= 10^4 copies/mL or > 2000 IU/mL), or acute or chronic active hepatitis C (hepatitis C virus [HCV] ribonucleic acid [RNA] >10^3 copies/mL), or simultaneously positive for HBsAg and HCV antibody
* History of gastrointestinal (GI) perforation and/or fistula within 6 months prior to the enrollment, excluding gastrostomy or enterostomy
* Interstitial lung disease requiring corticosteroids
* History of other primary malignant tumors, excluding:

  * Malignant tumors that achieved a complete response (CR) at least 2 years prior to enrollment and expected to require no treatment during the trial
  * Adequately treated nonmelanoma skin cancer or lentigo maligna with no sign of disease recurrence
  * Adequately treated carcinoma in situ with no sign of disease recurrence
  * Prostate, chronic lymphocytic leukemia (CLL) or other cancers where the indolent nature of tumor allows for and patient is cancer under active surveillance
* Pregnant or breastfeeding female subjects
* Acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may lead to the following consequences: increased investigational drug-related risks, interference with interpretation of trial results, or considered ineligible for participating in the trial by the investigators

  * If there are any uncertainties regarding the inclusion/exclusion, please contact the sponsor immediately and provide a complete medical history of the subject. The sponsor and principal investigator will discuss and determine the eligibility of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Progression-free rate | At 9 cycles (1 cycle = 21 days)
  Defined as the proportion of subjects with no confirmed progressive disease (PD) at 9 cycles assessed by the independent radiology review based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1) in the evaluable population.

SECONDARY OUTCOMES:
Duration of response | From first date of investigator-determined response to investigator-determined progressive disease (PD) or death in the subjects who have achieved complete response (CR) or partial response (PR), assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analyses of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Progression free survival | From treatment onset to either disease progression as defined by RECIST or death from any cause, or discontinuation of treatment for any reason, whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analyses of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Overall survival | From treatment onset to death, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analyses of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Objective response rate (complete response + partial response) | Up to 5 years
  Corresponding exact 95% confidence intervals (CIs) will be estimated using binomial distribution.
Stable disease rate | Up to 5 years
  Defined as stable disease for 9 cycles (1 cycle = 21 days). Corresponding exact 95% CIs will be estimated using binomial distribution.
Incidence of adverse events (AEs) | Up to 90 days after completion of treatment
  The incidence (frequency) of AEs, treatment-emergent (TE)AEs, treatment-related (TR)AEs, immunity related (ir)AEs, serious AEs, AEs resulting in treatment discontinuation, and AEs resulting in death will be summarized. The severity distribution of TEAEs, TRAEs, and irAEs will be summarized using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Ravi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT05026736/ICF_000.pdf